CLINICAL TRIAL: NCT03954145
Title: Comparison of Bonding Failure Rates of Fixed Mandibular Lingual Retainers in a French Sample Aged 11 or Older Comparing Prior Enamel Sandblasting With Conventional Pumice Polishing
Brief Title: Comparison of Bonding Failure Rates of Fixed Lingual Mandibular Retainers in a French Sample Aged 11 or Older, Comparing Prior Enamel Sandblasting With Conventional Pumice Polishing
Acronym: CONTORTHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 7434
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Detachment of Glued Mandibular Post-orthodontic Restraints

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PUMICING GROUP (Active Comparator): Lingual surfaces of the lower incisors and canines are pumiced before bonding the lingual retainer.
  Teeth are being cleaned using a brush loaded with pumice and mounted on a low speed contra-angle.Teeth are then etched and the multi-braided retainer wire is being bonded with composite onto the lingual surfaces of the lower canines and incisors
  Interventions: Procedure: Enamel pumicing before bonding the lingual retainer.
- SANDBLASTING GROUP (Experimental): Enamel is being initially prepared through sandblasting the lingual surfaces of the mandibular canines and incisors.
  Sandblasting is performed with the help of a MicroEtcher IIATM (Danville) which is projecting 50 μm Al2O3 particles onto the enamel surfaces. Teeth are subsequently etched and the retainer is then being bonded with composite onto the lingual surfaces of the mandibular incisors and canines.
  Interventions: Procedure: Enamel sandblasting before bonding the lingual retainer.

INTERVENTIONS:
Procedure: Enamel pumicing before bonding the lingual retainer. — Lingual surfaces of the lower incisors and canines are pumiced before bonding the lingual retainer.
  Teeth are being cleaned using a brush loaded with pumice and mounted on a low speed contra-angle. Teeth are then etched and the multi-braided retainer wire is being bonded with composite onto the lingual surfaces of the lower canines and incisors.
  Arms: PUMICING GROUP
Procedure: Enamel sandblasting before bonding the lingual retainer. — Enamel is being initially prepared through sandblasting the lingual surfaces of the mandibular canines and incisors.
  Sandblasting is performed with the help of a MicroEtcher IIATM (Danville) which is projecting 50 μm Al2O3 particles onto the enamel surfaces. Teeth are subsequently etched and the retainer is then being bonded with composite onto the lingual surfaces of the mandibular incisors and canines.
  Arms: SANDBLASTING GROUP

SUMMARY:
At the completion of orthodontic treatment, the position of the mandibular canines and incisors is being maintained on a routine basis by bonding a multi-braided wire retainer onto their lingual surfaces. One of the adverse events that might occur with time is the debonding of the wire from one or several lower anterior teeth . This event which can unfortunately get unnoticed by the patient can lead to unwanted tooth displacement. When the practionner detects such a debonding, he has to go through a laborious and lengthy procedure to rebond the wire. When on the other hand the patient notices himself such a debonding, he is to call in emergency his practitioner to get his retainer repaired. This leads to emergency visits that are susceptible to affect adversely his timetable. The prevalence of these bonding failures is estimated at 37% at 18 month follow-ups. It has been reported that with prior enamel sandblasting, bonding failure rate is reduced to 8% at 24 month follow-ups. However, no study has reported yet the debonding rate of lower fixed, comparing wires that have been bonded after prior enamel pumicing to those that were put in place after prior enamel sandblasting.

The expected result of this trial is a significantly decrease in bonding failure rate of mandibular lingual retainer when enamel surfaces are initially sandblasted compared to the ones which are pumiced. This reduction would lower the risk of unwanted tooth movement of mandibular incisors and canines after orthodontic treatment and decrease the number of emergency appointments for the patient and the practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 11 years of age
* At completion of fixed orthodontic therapy
* Presence of all 6 mandibular canines and incisors

Exclusion Criteria:

* Active decay
* Presence of dental restorations
* Tooth fracture
* Periodontal disease
* Structural anomalies affecting the lingual side of the mandibular incisors and canines
* Cleft lip and palate
* Cranio-facial syndrome
* Inability to obtain the patient informed consent

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Define the bonding failure rates of fixed mandibular lingual retainers during an 18 month follow-up, comparing prior enamel sandblasting with pumice polishing | Outcome is assessed with a probe and through visual examination at 3, 6, 9, 12, 15 and18 months after bonding the lingual retainer.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle de Médecine et Chirurgie Bucco-Dentaires, Strasbourg, Bas Rhin, France

REFERENCES:
- [Background] Kamm Q, Phonchareun E, Esquenet M, Rafflenbeul F, Severac F, Bolender Y. Comparison of bonding failure rates of mandibular retainers after 2 enamel preparations - sandblasting vs pumicing: An 18-month randomized controlled trial. Am J Orthod Dentofacial Orthop. 2025 Sep;168(3):262-272. doi: 10.1016/j.ajodo.2025.04.015. PMID 40885597